CLINICAL TRIAL: NCT02652065
Title: Cutaneous Microcirculation and Nervous Sensitivity in Psoriasis
Acronym: MicroPso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0425
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
Keywords: Psoriasis; Microcirculation; TRPV1
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy skin (Active Comparator): Local vasodilators (acetylcholine, sodium nitroprussiate and ppi water as control) will be delivered to patients by iontophoresis on healthy skin.
  The skin blood flow in response to these molecules will be followed by laser Doppler recordings.
  Interventions: Other: Acetylcholine iontophoresis; Other: Sodium Nitroprussiate iontophoresis; Other: ppi water iontophoresis; Other: Laser Doppler recording
- Psoriasis plaque (Experimental): Local vasodilators (acetylcholine, sodium nitroprussiate and ppi water as control) will be delivered to patients by iontophoresis on a psoriasis plaque (on the patient's back).
  The skin blood flow in response to these molecules will be followed by laser Doppler recordings.
  Interventions: Other: Acetylcholine iontophoresis; Other: Sodium Nitroprussiate iontophoresis; Other: ppi water iontophoresis; Other: Laser Doppler recording

INTERVENTIONS:
Other: Acetylcholine iontophoresis — Acetylcholine will be locally delivered to patients by iontophoresis successively on healthy skin and on psoriasis plaque (order determined by randomization).
Other: Sodium Nitroprussiate iontophoresis — Sodium Nitroprussiate will be locally delivered to patients by iontophoresis successively on healthy skin and on psoriasis plaque (order determined by randomization).
Other: ppi water iontophoresis — ppi water will be locally delivered to patients by iontophoresis successively on healthy skin and on psoriasis plaque (order determined by randomization).
Other: Laser Doppler recording — Skin blood flow will be recorded by laser Doppler during 2 minutes before iontophoresis, and during 30 minutes following iontophoretic delivery of vasodilators.

SUMMARY:
Psoriasis is a chronic inflammatory cutaneous disease, affecting 3% of the French population. Among psoriatic patients, 80% feel pain or cutaneous discomfort related to their pathology.

Neurogenic inflammation's role in psoriasis has recently been put forward by a study showing that TRPV1 ion channels are necessary to establish psoriasiform inflammation in mice.

The investigators hypothesize that there is a link between cutaneous sensory neuropathies and altered cutaneous microcirculation during psoriasis.

In order to test this hypothesis, local vasodilators will be delivered to patients by iontophoresis and their skin blood flow in response to these molecules will be followed by laser Doppler recordings. Two recordings will be performed for each patient, both on a psoriasis plaque and on uninvolved skin, in order for the patient to be his own internal control.

ELIGIBILITY:
Inclusion Criteria:

* Type I psoriasis
* Psoriasis plaques on the patient's back

Exclusion Criteria:

* BMI > 25
* Diabetic patient
* Arteriovenous disease history
* Ongoing anti-inflammatory treatment
* Major cardiovascular history (<3 months)
* Hypertension
* Topical treatment on the back skin (<7 days)
* Systemic treatment (steroids, methotrexate, retinoids, cyclosporine) or phototherapy (<1 month)
* Pregnant women
* Subject within exclusion period following a previous or ongoing biomedical study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
skin blood flow variation | at the latest 3 months after inclusion
  Skin blood flow variation on healthy skin and on psoriasis plaque will be measured by Laser Doppler in response to iontophoretic delivery of vasodilator substances (sodium nitroprussiate and acetylcholine) and ppi water. Skin blood flow will be recorded during 2 minutes before iontophoresis, and during 30 minutes following iontophoretic delivery of vasodilators.

SECONDARY OUTCOMES:
Sensory detection threshold | at the latest 3 months after inclusion
  Increasing size of Von Frey filaments will be placed onto patients' skin to assess sensory detection threshold.
Potential discomfort sensation thresholds | at the latest 3 months after inclusion
  Increasing size of Von Frey filaments will be placed onto patients' skin to assess potential discomfort sensation threshold.
Heat sensitivity | at the latest 3 months after inclusion
  Heat sensitivity will be assessed using hot (50°C) and cold (4°C) water

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot - Service de Dermatologie et Vénéréologie, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Le seuil de sensibilité tactile est augmenté sur les plaques de psoriasis comparée à celui des zones saines. Cette diminution de sensibilité tactile apparaît en absence de défaut de sensibilité sensorielle thermique ou vibratoire ou de discrimination tactile (test PIC/TOUCHE). L'exploration fonctionnelle de la microcirculation cutanée montre une perfusion fortement augmentée sur les plaques de psoriasis comparée à celle des zones saines. La microcirculation cutanée augmente en réponse à un chauffage local sur les 2 zones étudiées avec une amplitude plus marquée sur les plaques de psoriasis. La vasodilatation en réponse à l'application iontophorétique d'acétylcholine montre des résultats similaires. Ces réponses exacerbées pourraient être liées aux facteurs inflammatoires locaux, ce qui reste à démontrer dans le futur. - Conclusion : cette étude a permis de montrer des défauts de microcirculation cutanée sur les plaques de psoriasis, en l'absence de neuropathie sensorielle.